CLINICAL TRIAL: NCT00018863
Title: Methylphenidate Efficacy and Safety in ADHD Preschoolers
Brief Title: Treatment of Attention Deficit Hyperactivity Disorder in Preschool-Age Children (PATS)
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: New York State Psychiatric Institute (Other)
Collaborators: National Institute of Mental Health (NIMH) (NIH)
Responsible Party: Principal Investigator, Laurence Greenhill, Professor of Clinical Child and Adolescent Psychiatry, New York State Psychiatric Institute
Allocation: Randomized | Masking: Double | Purpose: Treatment
Other Study IDs: #3761; U01MH060903 (NIH); U01MH060642 (NIH); U01MH060943 (NIH); U01MH060848 (NIH); U01MH060900 (NIH); U01MH060833 (NIH); DSIR CT-M2
Record Dates: First submitted 2001-07-05; First posted 2001-07-09 (Estimated); Last update posted 2020-12-02 (Actual); Status verified 2020-11

CONDITIONS: Attention Deficit Disorder With Hyperactivity
Keywords: ADHD
MeSH Terms: conditions — Attention Deficit Disorder with Hyperactivity | interventions — Methylphenidate

INTERVENTIONS:
Drug: Methylphenidate

SUMMARY:
This research focuses on the treatment of Attention Deficit Hyperactivity Disorder (ADHD) in very young children. The medication being used is methylphenidate (Ritalin); it is being studied to determine its safety and how well it works to treat ADHD in preschool-age children (3-5.5 year olds).

DETAILED DESCRIPTION:
Young children age 3-5.5 years will be studied. The study includes treatment with different doses of methylphenidate and placebo; all children will receive active medication during the study. Prior to treatment, each child will receive a thorough psychiatric evaluation and each guardian will complete a 10-week workshop (2 hours/week). Throughout the study, parents and teachers will complete forms that report on the child's behavior and possible side effects. Participants will be monitored by regular visits with a study physician. Most participants will be involved in the study for up to 16 months to ensure optimal evaluation, dosing, and monitoring

ELIGIBILITY:
Boys and girls who are:

* Between the ages of 3-5.5 years
* Qualified as having ADHD by our diagnostic evaluations and clinical staff
* Otherwise generally healthy
* Willing, and have parents that are willing, to attend all visits required by the study
* Enrolled in some type of day-program: day care, preschool, nursery school, kindergarten, for at least 2 half days/week
* In classrooms with teachers that are willing to participate by completing rating scale

Ages: 3 Years to 5 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 165
Dates: Start 2001-04-01 (Actual); Primary Completion 2006-03-31 (Actual); Study Completion 2006-11-30 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Laurence Greenhill, M.D., Study Chair
Locations (6):
- United States (6):
  - University of California, Irvine, Irvine, California
  - University of California, Los Angeles, Los Angeles, California
  - Johns Hopkins University, Baltimore, Maryland
  - New York State Psychiatric Institute, New York, New York
  - New York University School of Medicine, New York, New York
  - Duke University Medical Center, Durham, North Carolina

REFERENCES:
- [Background] Schleifer M, Weiss G, Cohen N, Elman M, Cvejic H, Kruger E. Hyperactivity in preschoolers and the effect of methylphenidate. Am J Orthopsychiatry. 1975 Jan;45(1):38-50. doi: 10.1111/j.1939-0025.1975.tb01164.x. PMID 1089359
- [Background] Handen BL, Feldman HM, Lurier A, Murray PJ. Efficacy of methylphenidate among preschool children with developmental disabilities and ADHD. J Am Acad Child Adolesc Psychiatry. 1999 Jul;38(7):805-12. doi: 10.1097/00004583-199907000-00009. PMID 10405497
- [Background] Conners CK: Controlled trial of methylphenidate in preschool children with minimal brain dysfunction. Int J Ment Health (4):61-74, 1975.
- [Background] Barkley RA. The effects of methylphenidate on the interactions of preschool ADHD children with their mothers. J Am Acad Child Adolesc Psychiatry. 1988 May;27(3):336-41. doi: 10.1097/00004583-198805000-00012. No abstract available. PMID 3379016
- [Background] Mayes SD, Crites DL, Bixler EO, Humphrey FJ 2nd, Mattison RE. Methylphenidate and ADHD: influence of age, IQ and neurodevelopmental status. Dev Med Child Neurol. 1994 Dec;36(12):1099-107. doi: 10.1111/j.1469-8749.1994.tb11811.x. PMID 7525394
- [Background] Musten LM, Firestone P, Pisterman S, Bennett S, Mercer J. Effects of methylphenidate on preschool children with ADHD: cognitive and behavioral functions. J Am Acad Child Adolesc Psychiatry. 1997 Oct;36(10):1407-15. doi: 10.1097/00004583-199710000-00023. PMID 9334554
- [Result] Kollins S, Greenhill L, Swanson J, Wigal S, Abikoff H, McCRACKEN J, Riddle M, McGOUGH J, Vitiello B, Wigal T, Skrobala A, Posner K, Ghuman J, Davies M, Cunningham C, Bauzo A. Rationale, design, and methods of the Preschool ADHD Treatment Study (PATS). J Am Acad Child Adolesc Psychiatry. 2006 Nov;45(11):1275-1283. doi: 10.1097/01.chi.0000235074.86919.dc. PMID 17023869
- [Result] Swanson J, Greenhill L, Wigal T, Kollins S, Stehli A, Davies M, Chuang S, Vitiello B, Skrobala A, Posner K, Abikoff H, Oatis M, McCRACKEN J, McGOUGH J, Riddle M, Ghuman J, Cunningham C, Wigal S. Stimulant-related reductions of growth rates in the PATS. J Am Acad Child Adolesc Psychiatry. 2006 Nov;45(11):1304-1313. doi: 10.1097/01.chi.0000235075.25038.5a. PMID 17023868
- [Result] Greenhill L, Kollins S, Abikoff H, McCracken J, Riddle M, Swanson J, McGough J, Wigal S, Wigal T, Vitiello B, Skrobala A, Posner K, Ghuman J, Cunningham C, Davies M, Chuang S, Cooper T. Efficacy and safety of immediate-release methylphenidate treatment for preschoolers with ADHD. J Am Acad Child Adolesc Psychiatry. 2006 Nov;45(11):1284-1293. doi: 10.1097/01.chi.0000235077.32661.61. PMID 17023867
- [Result] McGOUGH J, McCRACKEN J, Swanson J, Riddle M, Kollins S, Greenhill L, Abikoff H, Davies M, Chuang S, Wigal T, Wigal S, Posner K, Skrobala A, Kastelic E, Ghuman J, Cunningham C, Shigawa S, Moyzis R, Vitiello B. Pharmacogenetics of methylphenidate response in preschoolers with ADHD. J Am Acad Child Adolesc Psychiatry. 2006 Nov;45(11):1314-1322. doi: 10.1097/01.chi.0000235083.40285.08. PMID 17023870
- [Result] Wigal T, Greenhill L, Chuang S, McGOUGH J, Vitiello B, Skrobala A, Swanson J, Wigal S, Abikoff H, Kollins S, McCRACKEN J, Riddle M, Posner K, Ghuman J, Davies M, Thorp B, Stehli A. Safety and tolerability of methylphenidate in preschool children with ADHD. J Am Acad Child Adolesc Psychiatry. 2006 Nov;45(11):1294-1303. doi: 10.1097/01.chi.0000235082.63156.27. PMID 17028508
- See also: Specific information on ADHD — http://www.nimh.nih.gov/health/topics/attention-deficit-hyperactivity-disorder-adhd/index.shtml